CLINICAL TRIAL: NCT05635032
Title: Host-microbiome Interactions in the Quest for Fibrosing ILD Biomarkers That Rule Acceleration
Brief Title: Fibrosing ILD Biomarkers That Rule Acceleration
Acronym: FIBRALUNG
Status: Recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Instituto de Investigação e Inovação em Saúde (i3S) (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Other Study IDs: FIBRALUNG
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Fibrosis; Sarcoidosis
MeSH Terms: conditions — Pulmonary Fibrosis; Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Creation of a biobank of peripheral blood (plasma, serum, DNA, RNA), bronchoalveolar lavage, pharyngeal swabs and lung tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IPF: Patients with Idiophatic Pulmonary Fibrosis (IPF), serving as a prototype of a progressive fibroproliferative disorder.
  Interventions: Other: Comprehensive clinical assessment and biological samples collection
- Progressive Pulmonary Fibrosis (non-IPF): Patients with non-IPF interstitial lung diseases, presenting a progressive fibrosing phenotype, or acute exacerbations.
  Interventions: Other: Comprehensive clinical assessment and biological samples collection
- Non-Progressive Pulmonary Fibrosis (non-IPF): Patients with fibrotic non-IPF interstitial lung diseases that are stable during a minimum follow-up of 24 months.
  Interventions: Other: Comprehensive clinical assessment and biological samples collection

INTERVENTIONS:
Other: Comprehensive clinical assessment and biological samples collection — To establish the first Portuguese registry and biobank of PF-ILDs, comprising both extensive patient-level data, and systematic biological sampling (DNA, RNA, plasma, serum, bronchoalveolar lavage, lung tissue) at baseline and repeated biological sampling of blood and pharyngeal swabs performed at 6, 12 and 18 months, or whenever progression criteria are met or an acute exacerbation occurs. Participants will have regular visits at maximum intervals of 6 months, when their clinical condition and lung function tests are reassessed. A high resolution computed tomography (HRCT) scan of the lung will be performed every 12 months. Progressive fibrosis will be diagnosed based on meeting at least two of the following three criteria, occurring within the last year: (i) worsening of symptoms; (ii) absolute decline in FVC ≥5% predicted or absolute decline in DLCO (corrected for Hb) ≥10% predicted; (iii) increased extent of fibrotic changes on HRCT.

SUMMARY:
FIBRALUNG is a prospective cohort study with biobank of samples from patients with pulmonary fibrosis, aiming to explore the molecular determinants of different clinical outcomes, acute exacerbations and mortality. We expect to gain deeper insight into fibroproliferative common pathways, particularly between idiopathic pulmonary fibrosis and fibrotic hypersensitivity pneumonitis, paving the way for new biomarkers that reflect the progressive phenotype, that eventually will support new targeted therapies.

Other idiopathic interstitial pneumonias, connective tissue disease-related interstitial lung diseases and sarcoidosis patients will be also recruited and their biological samples stored for further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-80 years
* People undergoing blood collection, lung biopsy and/or BAL as part of their diagnostic workup
* Willingness to undergo the follow-up protocol evaluations
* Treatment-naïve for disease-modifying drugs
* An HRCT scan performed within the last 12 months showing ≥10% fibrosis extent of the lungs

Exclusion Criteria:

* People who cannot give informed consent
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Interstitial Lung Diseases unit of Centro Hospitalar Universitário de São João (Porto, Portugal).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Discover biomarkers in progressive pulmonary fibrosis | 36 months
  Characterization of blood and tissue transcriptional signatures of progression and acute exacerbations, and validate findings at the protein expression level, which could be easily converted for clinical use as biomarkers.

SECONDARY OUTCOMES:
Change in microbiome profile in progressive pulmonary fibrosis | 24 months
  To assess the impact of microbiome features in clinical progression and higher risk of acute exacerbation

OTHER OUTCOMES:
Variation in Computed Tomography Lung Densitometry | 36 months
Proportion of patients varying FVC ⩾5% predicted within 1 year of follow-up | 36 months
Proportion of patients varying DLCO ⩾10% predicted within 1 year of follow-up | 36 months
Time to progression or exacerbation | 36 months
Survival | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Helder Novais Bastos, MD, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Centro Hospitalar Universitário São João, Porto, Portugal

REFERENCES:
- See also: Project presentation website — https://fibralung.pt/